CLINICAL TRIAL: NCT00909857
Title: A Multi-center, Double-blind, Double-dummy, Randomized, Controlled, Parallel-group Study to Assess Efficacy and Safety of SH T00658ID Compared to SH D593B in the Treatment of Primary Dysmenorrhea
Brief Title: Effect on Primary Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91781; 2008-005625-11 (EudraCT Number); 312042 (Other: Bayer)
Record Dates: First submitted 2009-04-24; First posted 2009-05-29 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Oral Contraception
MeSH Terms: interventions — Estradiol; dienogest; Ethinyl Estradiol; Levonorgestrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estradiol valerate, Dienogest (Natazia, Qlaira, BAY86-5027) (Experimental): Daily oral administration of one tablet SH T00658ID (BAY86-5027) plus one tablet placebo for 28 days without tablet-free interval for 3 treatment cycles
  Interventions: Drug: Estradiol valerate, Dienogest (Natazia, Qlaira, BAY86-5027); Drug: Placebo Match to SH T00658ID
- Ethinyl estradiol, Levonorgestrel (Miranova) (Active Comparator): Daily oral administration of one tablet placebo plus one tablet SH D593B (Miranova) for 28 days without tablet-free interval for 3 treatment cycles
  Interventions: Drug: Ethinyl estradiol, Levonorgestrel (Miranova); Drug: Placebo Match to SH D593B

INTERVENTIONS:
Drug: Estradiol valerate, Dienogest (Natazia, Qlaira, BAY86-5027) — Daily oral administration of one tablet SH T00658ID for 28 days per cycle in the respective treatment period; no tablet-free interval
  Arms: Estradiol valerate, Dienogest (Natazia, Qlaira, BAY86-5027)
Drug: Ethinyl estradiol, Levonorgestrel (Miranova) — Daily oral administration of one tablet for 28 days per cycle in the respective treatment period; no tablet-free interval
  Arms: Ethinyl estradiol, Levonorgestrel (Miranova)
Drug: Placebo Match to SH T00658ID — Daily oral administration of one tablet placebo for 28 days without tablet-free interval for 3 treatment cycles.
  Arms: Estradiol valerate, Dienogest (Natazia, Qlaira, BAY86-5027)
Drug: Placebo Match to SH D593B — Daily oral administration of one tablet placebo for 28 days without tablet-free interval for 3 treatment cycles.
  Arms: Ethinyl estradiol, Levonorgestrel (Miranova)

SUMMARY:
To investigate the potential benefits of a new oral contraceptive (SH T00658ID) on alleviating complaints of dysmenorrhea associated with oral contraceptive use.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy female subjects requesting contraception and suffering from primary dysmenorrhea with a sum score for dysmenorrheic pain intensity of >/= 8 over 2 baseline cycles documented by a prospective self-rated sum pain score
* Age: 14 - 50 years (inclusive; smokers must not be older than 30 years) at the time point of informed consent
* Normal cervical smear not requiring further follow-up (a cervical smear has to be taken at the screening visit, or a normal result has to be available that was documented within the last 6 months before the screening visit)
* Women with cyclic menstrual bleeding, defined by a cycle length between 25 and 35 days and no amenorrheic cycles or cycles without withdrawal bleeding during the last 3 months prior to visit 1.
* Able to tolerate ibuprofen and willing to use only Ibuprofen supplied for the study.

Exclusion Criteria:

* Pregnancy or lactation (delivery, abortion, or lactation within three cycles before the start of treatment)
* Obesity: body mass index (BMI) > 32 kg/m2
* Hypersensitivity to any of the study drug ingredients
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Presence or a history of venous or arterial thrombotic / thromboembolic events (e.g. deep venous thrombosis, pulmonary embolism, myocardial infarction) or of a cerebrovascular accident, including prodromi (e.g. transient ischemic attack, angina pectoris), and conditions that could increase the risk of suffering from any of the above mentioned disorders, e.g. a family history indicating a hereditary predispositionUndiagnosed abnormal genital bleeding
* Abuse of alcohol, drugs, or medicines (e.g. laxatives)
* Other contraceptive methods:

  * Sterilization
  * Oral, vaginal or transdermal hormonal contraception during treatment
  * Intra-uterine devices (IUD) with or without hormone release still in place within 30 days of visit 1
* Simultaneous participation in another clinical trial or participation in another clinical trial prior to study entry that might have an impact on the study objectives at the discretion of the investigator
* Major surgery scheduled for the study period

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 507 (Actual)
Dates: Start 2009-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (40):
- United States (10):
  - Tucson, Arizona
  - San Diego, California
  - Hialeah, Florida
  - Leesburg, Florida
  - Sandy Springs, Georgia
  - Idaho Falls, Idaho
  - Winston-Salem, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - La Crosse, Wisconsin
- Canada (5):
  - Langley, British Columbia
  - Toronto, Ontario
  - Pointe-Claire, Quebec
  - Ste-Foy, Quebec
  - Regina, Saskatchewan
- Chile (3):
  - Santiago
  - Talcahuano
  - Temuco
- Germany (7):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Hamburg, Hamburg
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Leipzig, Saxony
  - Bernburg, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
- Italy (10):
  - Francavilla Fontana, Brindisi
  - Bologna
  - Brescia
  - Milan
  - Modena
  - Perugia
  - Roma
  - Siena
  - Torino
  - Udine
- Philippines (5):
  - Cebu
  - Cebu City
  - Davao City
  - Metro Manila
  - Quezon City

REFERENCES:
- [Derived] Schroll JB, Black AY, Farquhar C, Chen I. Combined oral contraceptive pill for primary dysmenorrhoea. Cochrane Database Syst Rev. 2023 Jul 31;7(7):CD002120. doi: 10.1002/14651858.CD002120.pub4. PMID 37523477
- [Derived] Petraglia F, Parke S, Serrani M, Mellinger U, Romer T. Estradiol valerate plus dienogest versus ethinylestradiol plus levonorgestrel for the treatment of primary dysmenorrhea. Int J Gynaecol Obstet. 2014 Jun;125(3):270-4. doi: 10.1016/j.ijgo.2013.11.017. Epub 2014 Mar 11. PMID 24713413
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged 14 to 50 years with a need for oral contraception suffering from primary dysmenorrhea were recruited at specialized study sites.
Pre-assignment Details: Out of 771 participants screened, 264 failed screening, mostly due to not meeting in-/exclusion criteria (155), withdrawal of consent (49), loss to follow-up (36) or pregnancy (10). Thus, 507 participants were randomized (253 to Estradiol valerate/Dienogest and 254 to Ethinyl estradiol/Levonorgestrel).
Period: Overall Study
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Started | 253 | 254
Treated | 234 | 230
Completed | 217 | 209
Not Completed | 36 | 45
Not completed — Withdrawal by Subject | 6 | 10
Not completed — Adverse Event | 5 | 5
Not completed — Lost to Follow-up | 2 | 5
Not completed — Protocol Violation | 2 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Other | 1 | 0
Not completed — Did not receive study medication | 19 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova) | Total
Number analyzed (Participants) | 234 | 230 | 464
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (7.9) | 27.6 (8.0) | 27.8 (7.9)
Age, Customized [Number; unit: Participants]
  less than 18 years of age | 11 | 13 | 24
  18 years of age or older | 223 | 217 | 440
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 230 | 464
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change Between Baseline Evaluation Period and Treatment Evaluation Period in the Number of Days With Dysmenorrheic Pain
Description: Dysmenorrheic pain was defined as pelvic pain during the menstrual/withdrawal bleeding episode and the 2 days before this episode. Baseline period: 2 days before the first menstrual bleeding until 3rd day before the 3rd menstrual bleeding (normalized to a standard 56-day period). Treatment period: 2 days before the withdrawal bleeding (WB) of the 1st evaluable treatment cycle until 3rd day before the WB of the cycle after the 2nd evaluable treatment cycle (normalized to a standard 56-day period).
Time Frame: baseline period (2 baseline cycles, usually 56 days) vs. treatment period (on-treatment cycles 2 and 3, usually 56 days)
Population: Full analysis set (FAS): all subjects admitted to the treatment phase who took at least 1 tablet of study medication or comparator, and for whom at least 1 observation after admission to treatment was available, all participants with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 225 | 219
Days | -4.6 (4.6) | -4.2 (4.2)

2. Secondary Outcome: Change Between Baseline Evaluation Period and Treatment Evaluation Period in the Sum of Score Points of Dysmenorrheic Pain
Description: Dysmenorrheic pain: pelvic pain during menstrual/withdrawal bleeding (WB) episode and 2 days before. Scores per day: 0 No pain; 1 Mild pain with no need for painkiller; 2 Moderate pain with need for painkiller; 3 Severe pain with need for painkiller. Baseline period: 2 days before 1st menstrual bleeding until 3rd day before 3rd menstrual bleeding (normalized to standard 56-day period). Treatment period: 2 days before WB of 1st treatment cycle until 3rd day before WB of the cycle after 2nd treatment cycle (normalized to standard 56-day period). Score difference min -168 (best), max 168 (worst)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 225 | 219
Scores on a scale | -10.6 (9.7) | -10.0 (8.9)

3. Secondary Outcome: Change Between Baseline Evaluation Period and Treatment Evaluation Period in Number of Days With Pelvic Pain Independent of Occurrence of Vaginal Bleeding
Description: Baseline period: 2 days before the first menstrual bleeding until 3rd day before the 3rd menstrual bleeding (normalized to a standard 56-day period). Treatment period: 2 days before the withdrawal bleeding (WB) of the 1st evaluable treatment cycle until 3rd day before the WB of the cycle after the 2nd evaluable treatment cycle (normalized to a standard 56-day period).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 225 | 219
Days | -4.0 (5.7) | -3.7 (5.7)

4. Secondary Outcome: Change Between Baseline Evaluation Period and Treatment Evaluation Period in Number of Days With Pelvic Pain During Unscheduled Bleeding
Description: Evaluated was the number of days with bleeding-associated pelvic pain, excluding days during withdrawal bleeding (WB) and the 2 days preceding such WB, and during administration deviation bleeding and the 2 days preceding such bleeding (normalized to a standard 56-day period). Baseline period: 2 days before first menstrual bleeding until 3rd day before 3rd menstrual bleeding (normalized to standard 56-day period). Treatment period: 2 days before WB of the 1st treatment cycle until 3rd day before the WB of the cycle after the 2nd treatment cycle (normalized to standard 56-day period).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 225 | 219
Days | 0.3 (2.6) | 0.1 (2.0)

5. Secondary Outcome: Change Between Baseline Evaluation Period and Treatment Evaluation Period in Rescue Medication Use (Only Bleeding Episodes Used Including the Two Days Before the Episode)
Description: Rescue medication use was standardized intake of 200 mg Ibuprofen tablets. Baseline period: 2 days before the first menstrual bleeding until 3rd day before the 3rd menstrual bleeding (normalized to a standard 56-day period). Treatment period: 2 days before the withdrawal bleeding (WB) of the 1st evaluable treatment cycle until 3rd day before the WB of the cycle after the 2nd evaluable treatment cycle (normalized to a standard 56-day period).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tablets
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 225 | 219
Tablets | -6.2 (14.8) | -6.6 (12.3)

6. Secondary Outcome: Change Between Baseline Evaluation Period and Treatment Evaluation Period in Rescue Medication Use (Entire Evaluation Period Used)
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tablets
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 225 | 219
Tablets | -4.5 (19.9) | -5.6 (14.3)

7. Secondary Outcome: Percentage of Participants With Interference of Dysmenorrheic Pain With Work/School and Social or Other Activity (Only Bleeding Episodes Used Including the Two Days Before)
Description: Interference of dysmenorrheic pain with work/school and social or other activity was assessed (yes/no). Baseline period: 2 days before the first menstrual bleeding until 3rd day before the 3rd menstrual bleeding (normalized to a standard 56-day period). Treatment period: 2 days before the withdrawal bleeding (WB) of the 1st evaluable treatment cycle until 3rd day before the WB of the cycle after the 2nd evaluable treatment cycle (normalized to a standard 56-day period).
Time Frame: as for outcome 1
Population: Full analysis set (FAS): all subjects admitted to the treatment phase who took at least 1 tablet of study medication or comparator, and for whom at least 1 observation after admission to treatment was available
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 230
Percentage of participants
  Baseline period-daily activities impaired | 92.3 | 91.3
  Baseline period- leisure activities impaired | 90.6 | 89.6
  Treatment period-daily activities impaired | 51.7 | 56.5
  Treatment period- leisure activities impaired | 47.9 | 56.5

8. Secondary Outcome: Percentage of Participants With Interference of Dysmenorrheic Pain With Work/School and Social or Other Activity (Entire Evaluation Period Used)
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 230
Percentage of Participants
  Baseline period-daily activities impaired | 93.2 | 92.2
  Baseline period- leisure activities impaired | 92.3 | 90.0
  Treatment period-daily activities impaired | 54.7 | 60.0
  Treatment period- leisure activities impaired | 52.6 | 61.3

9. Secondary Outcome: Percentage of Participants Satisfied With Study Treatment
Description: Participants were asked to express the degree of their satisfaction with study treatment.
Time Frame: From cycle 1 to cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 225 | 216
Percentage of participants
  Missing | 0.9 | 1.3
  Very satisfied | 53.4 | 50.4
  Saatisfied | 32.1 | 30.0
  Neither satisfied nor dissatisfied | 7.3 | 8.3
  Dissatisfied | 2.1 | 3.5
  Very dissatisfied | 0.4 | 0.4

10. Secondary Outcome: Number of Days With Bleeding or Spotting
Description: Bleeding/spotting episodes (day[s] with bleeding/spotting preceded and followed by at least 2 bleeding/spotting-free days) were described using the reference period (RP) method (length of RP: 90 days) recommended by the World Health Organization. 1st RP started on the 1st day of study medication. The total number of days during bleeding or spotting episodes was counted. Spotting = less than associated with normal menstruation relative to the subject's experience with no need for sanitary protection (except for panty liners). Bleeding = any bleeding of greater intensity than spotting.
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 201 | 197
Days | 20.0 (8.8) | 23.6 (9.7)

11. Secondary Outcome: Number of Episodes With Bleeding or Spotting
Description: as for outcome 10
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 201 | 197
Episodes | 3.9 (1.0) | 4.1 (0.8)

12. Secondary Outcome: Mean Length of Bleeding or Spotting Episodes
Description: as for outcome 10
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 201 | 197
Days | 5.17 (2.26) | 5.83 (2.35)

13. Secondary Outcome: Maximum Length of Bleeding or Spotting Episodes
Description: as for outcome 10
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 201 | 197
Days | 7.1 (3.8) | 8.4 (5.6)

14. Secondary Outcome: Difference in Duration Between Longest and Shortest Bleeding or Spotting Episode
Description: as for outcome 10
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 201 | 197
Days | 3.6 (3.6) | 4.6 (5.6)

15. Secondary Outcome: Number of Days With Spotting-only
Description: as for outcome 10
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 201 | 197
Days | 7.3 (6.9) | 7.6 (7.5)

16. Secondary Outcome: Number of Episodes With Spotting-only
Description: as for outcome 10
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 201 | 197
Episodes | 0.5 (0.8) | 0.4 (0.7)

17. Secondary Outcome: Mean Length of Spotting Only Episodes
Description: as for outcome 10
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 67 | 51
Days | 3.29 (2.39) | 3.26 (2.79)

18. Secondary Outcome: Maximum Length of Spotting Only Episodes
Description: as for outcome 10
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 67 | 51
Days | 3.9 (3.1) | 3.6 (3.0)

19. Secondary Outcome: Difference in Duration Between Longest and Shortest Spotting Only Episode
Description: as for outcome 10
Time Frame: From day 1 to day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 67 | 51
Days | 1.2 (2.5) | 0.7 (1.5)

20. Secondary Outcome: Percentage of Participants With Withdrawal Bleeding at Cycle 1
Description: Withdrawal bleeding was defined as the first bleeding episode after complete or partial progestogen withdrawal (i.e. the first episode starting after the last day of progestogen intake). If a bleeding episode was ongoing on the last day of progestogen intake and the following day, this episode was regarded as the withdrawal bleeding episode, as long as it had started not more than 4 days before the progestogen withdrawal.
Time Frame: At cycle 1 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 222
Percentage of Participants | 91.2 | 93.2

21. Secondary Outcome: Percentage of Participants With Withdrawal Bleeding at Cycle 3
Description: as for outcome 20
Time Frame: At cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 204 | 198
Percentage of Participants | 68.1 | 79.3

22. Secondary Outcome: Length of Withdrawal Bleeding Episodes at Cycle 1
Description: as for outcome 20
Time Frame: At cycle 1 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 206 | 207
Days | 5.2 (2.7) | 5.4 (2.4)

23. Secondary Outcome: Length of Withdrawal Bleeding Episodes at Cycle 3
Description: as for outcome 20
Time Frame: At cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 139 | 157
Days | 4.5 (1.7) | 5.2 (2.0)

24. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 1
Description: Withdrawal bleeding was defined as the first bleeding episode after complete or partial progestogen withdrawal (i.e. the first episode starting after the last day of progestogen intake). If a bleeding episode was ongoing on the last day of progestogen intake and the following day, this episode was regarded as the withdrawal bleeding episode, as long as it had started not more than 4 days before the progestogen withdrawal. Intensity was defined as: 1 = none, 2 = spotting, 3 = light, 4 = normal, 5 = heavy.
Time Frame: At cycle 1 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 206 | 207
Scores on a scale | 3.7 (1.0) | 4.0 (0.9)

25. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 3
Description: as for outcome 24
Time Frame: At cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 139 | 157
Scores on a scale | 3.7 (0.8) | 4.1 (0.8)

26. Secondary Outcome: Onset of Withdrawal Bleeding Episodes at Cycle 1
Description: as for outcome 20
Time Frame: At cycle 1 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 206 | 207
Days | 4.8 (7.0) | 4.9 (5.9)

27. Secondary Outcome: Onset of Withdrawal Bleeding Episodes at Cycle 3
Description: as for outcome 20
Time Frame: At cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 139 | 157
Days | 3.1 (3.7) | 4.3 (4.4)

28. Secondary Outcome: Percentage of Participants With Intracyclic Bleeding at Cycle 1
Description: Intracyclic bleeding episodes were any bleeding episodes not qualifying as withdrawal bleeding. The latter was defined as the first bleeding episode after complete or partial progestogen withdrawal (i.e. the first episode starting after the last day of progestogen intake). If a bleeding episode was ongoing on the last day of progestogen intake and the following day, this episode was regarded as the withdrawal bleeding episode, as long as it had started not more than 4 days before the progestogen withdrawal.
Time Frame: At cycle 1 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 222
Percentage of Participants | 19.0 | 16.7

29. Secondary Outcome: Percentage of Participants With Intracyclic Bleeding at Cycle 3
Description: as for outcome 28
Time Frame: At cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 204 | 198
Percentage of Participants | 10.8 | 11.6

30. Secondary Outcome: Number of Intracyclic Bleeding Episodes at Cycle 1
Description: as for outcome 28
Time Frame: At cycle 1 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 222
Episodes | 0.2 (0.5) | 0.2 (0.4)

31. Secondary Outcome: Number of Intracyclic Bleeding Episodes at Cycle 3
Description: as for outcome 28
Time Frame: At cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 204 | 198
Episodes | 0.1 (0.3) | 0.1 (0.4)

32. Secondary Outcome: Maximum Length of Intracyclic Bleeding Episodes at Cycle 1
Description: as for outcome 28
Time Frame: At cycle 1 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 43 | 37
Days | 6.0 (5.4) | 6.2 (5.7)

33. Secondary Outcome: Maximum Length of Intracyclic Bleeding Episodes at Cycle 3
Description: as for outcome 28
Time Frame: At cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 22 | 23
Days | 5.5 (4.7) | 4.9 (4.1)

34. Secondary Outcome: Number of Intracyclic Bleeding Days at Cycle 1
Description: Intracyclic bleeding episodes were any bleeding episodes not qualifying as withdrawal bleeding. The latter was defined as the first bleeding episode after complete or partial progestogen withdrawal (i.e. the first episode starting after the last day of progestogen intake). If a bleeding episode was ongoing on the last day of progestogen intake and the following day, this episode was regarded as the withdrawal bleeding episode, as long as it had started not more than 4 days before the progestogen withdrawal. The total number of days during intracyclic bleeding episodes was counted.
Time Frame: At cycle 1 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 222
Days | 1.2 (3.5) | 1.0 (3.3)

35. Secondary Outcome: Number of Intracyclic Bleeding Days at Cycle 3
Description: as for outcome 34
Time Frame: At cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 204 | 198
Days | 0.6 (2.3) | 0.6 (2.1)

36. Secondary Outcome: Percentage of Participants With Maximum Intensity of Intracyclic Bleeding Episodes at Cycle 1
Description: Intracyclic bleeding episodes were any bleeding episodes not qualifying as withdrawal bleeding. The latter was defined as the first bleeding episode after complete or partial progestogen withdrawal (i.e. the first episode starting after the last day of progestogen intake). If a bleeding episode was ongoing on the last day of progestogen intake and the following day, this episode was regarded as the withdrawal bleeding episode, as long as it had started not more than 4 days before the progestogen withdrawal. Intensity could be described as spotting, light, normal or heavy.
Time Frame: At cycle 1 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 43 | 37
Percentage of participants
  Spotting | 53.5 | 62.2
  Light | 30.2 | 10.8
  Normal | 9.3 | 13.5
  Heavy | 7.0 | 13.5

37. Secondary Outcome: Percentage of Participants With Maximum Intensity of Intracyclic Bleeding Episodes at Cycle 3
Description: as for outcome 36
Time Frame: At cycle 3 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 22 | 23
Percentage of participants
  Spotting | 45.5 | 30.4
  Light | 27.3 | 21.7
  Normal | 13.6 | 30.4
  Heavy | 13.6 | 17.4

38. Secondary Outcome: Percentage of Participants Missing Time From Work Due to Dysmenorrheic Pain at Screening
Description: The investigator was asked to interview the participant and record the number of missed hours/days from work due to dysmenorrheic pain in the previous menstrual cycle.
Time Frame: At screening (28 days)
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 230
Percentage of Participants
  Missing | 0.4 | 0.0
  Never | 38.0 | 40.4
  4 working hours | 16.2 | 16.1
  1 working day | 26.5 | 29.6
  >= 2 working days | 18.8 | 13.9

39. Secondary Outcome: Percentage of Participants Missing Time From Work Due to Dysmenorrheic Pain at Baseline Cycle
Description: as for outcome 38
Time Frame: At Baseline (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 229
Percentage of Participants
  Missing | 0.0 | 0.0
  Never | 47.9 | 51.7
  4 working hours | 13.2 | 11.7
  1 working day | 20.9 | 23.9
  >= 2 working days | 17.9 | 12.2

40. Secondary Outcome: Percentage of Participants Missing Time From Work Due to Dysmenorrheic Pain at Cycle 2
Description: as for outcome 38
Time Frame: At cycle 2 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 224 | 212
Percentage of Participants
  Missing | 0.0 | 0.0
  Never | 78.6 | 72.6
  4 working hours | 8.5 | 6.5
  1 working day | 6.4 | 8.7
  >= 2 working days | 2.1 | 4.3

41. Secondary Outcome: Percentage of Participants Missing Time From Work Due to Dysmenorrheic Pain at Final Examination
Description: as for outcome 38
Time Frame: At final examination (28 days)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 217
Percentage of Participants
  Missing | 0.4 | 0.0
  Never | 85.9 | 85.2
  4 working hours | 5.6 | 2.6
  1 working day | 3.0 | 4.8
  >= 2 working days | 1.7 | 1.7

42. Secondary Outcome: Own Costs of Physiotherapy Per Treatment Converted to U.S. Dollars as Measured by Resource Use Questionnaire
Description: The participants were asked to complete a resource use questionnaire indicating their own costs of physiotherapy per treatment of dysmenorrheic pain. Costs were converted to U.S. dollars.
Time Frame: At screening (average over 3 months before screening)
Population: as for outcome 1
Measure: Median (Full Range); unit: Dollars
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 173 | 174
Dollars | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

43. Secondary Outcome: Own Costs of Pain Medication Per Treatment Converted to U.S. Dollars as Measured by Resource Use Questionnaire
Description: The participants were asked to complete a resource use questionnaire indicating their own costs of pain medication per treatment of dysmenorrheic pain. Costs were converted to U.S. dollars.
Time Frame: At screening (average over 3 months before screening)
Population: as for outcome 1
Measure: Median (Full Range); unit: Dollars
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 206 | 195
Dollars | 5.46 [0.00 to 30.00] | 5.04 [0.00 to 27.49]

44. Secondary Outcome: Own Costs of Vitamins Per Treatment Converted to U.S. Dollars as Measured by Resource Use Questionnaire
Description: The participants were asked to complete a resource use questionnaire indicating their own costs of vitamins per treatment of dysmenorrheic pain. Costs were converted to U.S. dollars.
Time Frame: At screening (average over 3 months before screening)
Population: as for outcome 1
Measure: Median (Full Range); unit: Dollars
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 173 | 176
Dollars | 0.00 [0.00 to 65.45] | 0.00 [0.00 to 65.45]

45. Secondary Outcome: Own Costs of Massages Per Treatment Converted to U.S. Dollars as Measured by Resource Use Questionnaire
Description: The participants were asked to complete a resource use questionnaire indicating their own costs of massages per treatment of dysmenorrheic pain. Costs were converted to U.S. dollars.
Time Frame: At screening (average over 3 months before screening)
Population: as for outcome 1
Measure: Median (Full Range); unit: Dollars
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 172 | 172
Dollars | 0.00 [0.00 to 60.00] | 0.00 [0.00 to 295.98]

46. Secondary Outcome: Own Costs of Acupuncture Per Treatment Converted to U.S. Dollars as Measured by Resource Use Questionnaire
Description: The participants were asked to complete a resource use questionnaire indicating their own costs of acupuncture per treatment of dysmenorrheic pain. Costs were converted to U.S. dollars.
Time Frame: At screening (average over 3 months before screening)
Population: as for outcome 1
Measure: Median (Full Range); unit: Dollars
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 174 | 174
Dollars | 0.00 [0.00 to 150.00] | 0.00 [0.00 to 74.00]

47. Secondary Outcome: Own Costs of Medical Counseling Per Treatment Converted to U.S. Dollars as Measured by Resource Use Questionnaire
Description: The participants were asked to complete a resource use questionnaire indicating their own costs of medical counseling per treatment of dysmenorrheic pain. Costs were converted to U.S. dollars.
Time Frame: At screening (average over 3 months before screening)
Population: as for outcome 1
Measure: Median (Full Range); unit: Dollars
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 170 | 170
Dollars | 0.00 [0.00 to 271.68] | 0.00 [0.00 to 98.17]

48. Secondary Outcome: Own Costs of Alternative Medicine Per Treatment Converted to U.S. Dollars as Measured by Resource Use Questionnaire
Description: The participants were asked to complete a resource use questionnaire indicating their own costs of alternative medicine per treatment of dysmenorrheic pain. Costs were converted to U.S. dollars.
Time Frame: At screening (average over 3 months before screening)
Population: as for outcome 1
Measure: Median (Full Range); unit: Dollars
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 177 | 175
Dollars | 0.00 [0.00 to 196.34] | 0.00 [0.00 to 110.00]

49. Secondary Outcome: Own Costs of Herbs/Teas Per Treatment Converted to U.S. Dollars as Measured by Resource Use Questionnaire
Description: The participants were asked to complete a resource use questionnaire indicating their own costs of herbs/teas per treatment of dysmenorrheic pain. Costs were converted to U.S. dollars.
Time Frame: At screening (average over 3 months before screening)
Population: as for outcome 1
Measure: Median (Full Range); unit: Dollars
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 183 | 179
Dollars | 0.00 [0.00 to 30.00] | 0.00 [0.00 to 10.00]

50. Secondary Outcome: Other Own Costs Per Treatment Converted to U.S. Dollars as Measured by Resource Use Questionnaire
Description: The participants were asked to complete a resource use questionnaire indicating their other own costs per treatment of dysmenorrheic pain. Costs were converted to U.S. dollars.
Time Frame: At screening (average over 3 months before screening)
Population: as for outcome 1
Measure: Median (Full Range); unit: Dollars
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 192 | 194
Dollars | 0.00 [0.00 to 15.00] | 0.00 [0.00 to 42.00]

51. Secondary Outcome: Participants With Improvement in the Investigators' Assessment in the Clinical Global Impression
Description: The Clinical Global Impression Scale (CGI) is a widely used rating scale/assessment instrument in psychopharmacology research in general, and in studies on women's health in particular. Investigators were asked to rate the participants' improvement during the course of the study.
Time Frame: At cycle 2 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 223 | 210
Participants
  Missing | 0 | 0
  Not assessed | 1 | 1
  Very much improved | 63 | 42
  Much improved | 87 | 84
  Minimally improved | 49 | 54
  No change | 17 | 23
  Minimally worse | 6 | 3
  Much worse | 0 | 6

52. Secondary Outcome: Participants With Improvement in Participants' Assessment in the Clinical Global Impression
Description: The Clinical Global Impression Scale (CGI) is a widely used rating scale/assessment instrument in psychopharmacology research in general, and in studies on women's health in particular. Participants were asked to rate their improvement during the course of the study.
Time Frame: At cycle 2 (28 days per cycle)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 223 | 210
Participants
  Missing | 1 | 0
  Not assessed | 1 | 1
  Very much improved | 60 | 46
  Much improved | 91 | 75
  Minimally improved | 47 | 57
  No change | 18 | 24
  Minimally worse | 5 | 4
  Much worse | 0 | 3

53. Secondary Outcome: Physical Functioning as Measured by General Health and Well-being Questionnaire SF-36 at Baseline Cycle
Description: The standard questionnaire SF-36v1, a general health status measure used to evaluate patient populations and to compare health status across different populations, was completed by participants as a self-administered native language version. Percentages of absolute scores were calculated such that 0 represents the lowest possible score (worst outcome) and 100 the highest possible score (best outcome)
Time Frame: At baseline cycle (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 229
Scores on a scale | 90.2 (16.7) | 89.6 (17.5)

54. Secondary Outcome: Physical Functioning as Measured by General Health and Well-being Questionnaire SF-36 at Final Examination
Description: as for outcome 53
Time Frame: at final examination (28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 217
Scores on a scale | 93.7 (14.2) | 92.5 (15.0)

55. Secondary Outcome: Social Functioning as Measured by General Health and Well-being Questionnaire SF-36 at Baseline Cycle
Description: as for outcome 53
Time Frame: At baseline cycle (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 229
Scores on a scale | 78.85 (18.99) | 77.35 (20.56)

56. Secondary Outcome: Social Functioning as Measured by General Health and Well-being Questionnaire SF-36 at Final Examination
Description: as for outcome 53
Time Frame: At final examination (28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 217
Scores on a scale | 85.95 (19.09) | 84.79 (17.36)

57. Secondary Outcome: Mental Health as Measured by General Health and Well-being Questionnaire SF-36 at Baseline Cycle
Description: as for outcome 53
Time Frame: At baseline cycle (28 days per cycle)
Population: Full analysis set (FAS): all subjects admitted to the treatment phase who took at least 1 tablet of study medication or comparator, and for whom at least 1 observation after admission to treatment was available, all participants wit assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 229
Scores on a scale | 73.6 (15.6) | 72.6 (16.3)

58. Secondary Outcome: Mental Health as Measured by General Health and Well-being Questionnaire SF-36 at Final Examination
Description: as for outcome 53
Time Frame: At final examination (28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 217
Scores on a scale | 77.3 (14.9) | 76.4 (14.7)

59. Secondary Outcome: Vitality as Measured by General Health and Well-being Questionnaire SF-36 at Baseline Cycle
Description: as for outcome 53
Time Frame: At baseline cycle (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 229
Scores on a scale | 62.6 (18.0) | 62.2 (18.2)

60. Secondary Outcome: Vitality as Measured by General Health and Well-being Questionnaire SF-36 at Final Examination
Description: as for outcome 53
Time Frame: At final examination (28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 217
Scores on a scale | 68.2 (17.0) | 67.2 (16.8)

61. Secondary Outcome: General Health as Measured by General Health and Well-being Questionnaire SF-36 at Baseline Cycle
Description: as for outcome 53
Time Frame: At baseline cycle (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 229
Scores on a scale | 75.8 (17.5) | 72.7 (16.9)

62. Secondary Outcome: General Health as Measured by General Health and Well-being Questionnaire SF-36 at Final Examination
Description: as for outcome 53
Time Frame: At final examination (28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 217
Scores on a scale | 77.2 (17.9) | 76.5 (16.6)

63. Secondary Outcome: Role Physical as Measured by General Health and Well-being Questionnaire SF-36 at Baseline Cycle
Description: as for outcome 53
Time Frame: At baseline cycle (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 229
Scores on a scale | 77.8 (33.6) | 79.4 (32.7)

64. Secondary Outcome: Role Physical as Measured by General Health and Well-being Questionnaire SF-36 at Final Examination
Description: as for outcome 53
Time Frame: At final examination (28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 217
Scores on a scale | 89.6 (23.0) | 87.9 (25.9)

65. Secondary Outcome: Role Emotional as Measured by General Health and Well-being Questionnaire SF-36 at Baseline Cycle
Description: as for outcome 53
Time Frame: At baseline cycle (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 229
Scores on a scale | 81.91 (31.50) | 79.18 (34.74)

66. Secondary Outcome: Role Emotional as Measured by General Health and Well-being Questionnaire SF-36 at Final Examination
Description: as for outcome 53
Time Frame: At final examination (28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 217
Scores on a scale | 88.64 (26.36) | 83.87 (30.28)

67. Secondary Outcome: Bodily Pain as Measured by General Health and Well-being Questionnaire SF-36 at Baseline Cycle
Description: as for outcome 53
Time Frame: At baseline cycle (28 days per cycle)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 234 | 229
Scores on a scale | 50.7 (24.4) | 51.8 (23.0)

68. Secondary Outcome: Bodily Pain as Measured by General Health and Well-being Questionnaire SF-36 at Final Examination
Description: as for outcome 53
Time Frame: At final examination (28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Number analyzed (Participants) | 226 | 217
Scores on a scale | 77.0 (21.5) | 74.0 (22.1)

ADVERSE EVENTS:
Arm/Group | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) | Ethinyl Estradiol, Levonorgestrel (Miranova)
Serious Adverse Events (participants affected / at risk) | 2/234 | 2/230
Other Adverse Events (participants affected / at risk) | 131/234 | 122/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) (N=234) | Ethinyl Estradiol, Levonorgestrel (Miranova) (N=230)
Helminthic infection (Infections and infestations) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Ovarian torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Valerate, Dienogest (Natazia, Qlaira, BAY86-5027) (N=234) | Ethinyl Estradiol, Levonorgestrel (Miranova) (N=230)
Dental caries (Gastrointestinal disorders) | 5 (10) | 2 (7)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (6)
Inflammation (General disorders) | 7 (7) | 3 (3)
Influenza (Infections and infestations) | 2 (2) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 7 (10)
Headache (Nervous system disorders) | 32 (55) | 34 (55)
Tension headache (Nervous system disorders) | 14 (40) | 9 (43)
Cervical dysplasia (Reproductive system and breast disorders) | 7 (7) | 9 (9)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 3 (4) | 5 (6)
Dysmenorrhoea (Reproductive system and breast disorders) | 87 (208) | 82 (210)
Metrorrhagia (Reproductive system and breast disorders) | 18 (28) | 13 (17)
Cervix inflammation (Reproductive system and breast disorders) | 9 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days